CLINICAL TRIAL: NCT01944748
Title: Family Mediation Program For At-Risk Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA031910 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-18 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Family Functioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Mediation (Experimental): Families receive FARS family mediation program after completing baseline survey.
  Interventions: Behavioral: Families Able To Resolve Situations (FARS)
- Wait-list control (No Intervention): Families receive FARS family mediation program after completing baseline, 6-week and 12-week surveys.

INTERVENTIONS:
Behavioral: Families Able To Resolve Situations (FARS) — Family mediation is a method of resolving conflicts between parents and teens. During the mediation session, the parent and teen each meet one-on-one with a trained volunteer mediator, who is a neutral person who listens to each party's concerns without taking sides. Then the parent and teen come together and meet with this mediator to work on resolving conflicts they are having. Families participate in up to 3 mediation sessions.
  Arms: Family Mediation

SUMMARY:
The goal of this project is to conduct a pilot evaluation of a parent-child mediation program for at-risk youth. It is investigating whether families who receive parent-child mediation show greater improvement in family functioning, as well as adolescent substance use, academic performance, and delinquency, over a 6-week and 12-week period compared to a wait-list control sample.

ELIGIBILITY:
Inclusion Criteria:

1. Has a child referred to FARS due to having problems in any of the following areas: (a) poor grades; (b) truancy; (c) defiant behavior; (d) running away; (e) delinquency; (f) substance use
2. Agrees to participate in at least one FARS mediation session
3. Agrees to complete 3 surveys and be available over the next 3 months for follow-up
4. Fluent in English or Spanish

   -

   Exclusion Criteria: Families referred to FARS due to: (a) conflicts involving gang violence (e.g., shootings, killings); (b) conflicts involving weapons; (c) arson; (d) conflicts involving explicit sex activities; (e) conflicts involving domestic violence/child abuse; and (f) threats to harm self or others.

   -

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2011-07; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Positive Family Relations | 6-week
  6-item Positive Family Relations measure adapted from the Cohesion subscale of Moos & Moos Family Environment Scale (Metzler et al., 1998; Journal of Family Psychology, 12, 600-619). Items are rated on a 5-point scale ("not at all" to "very much") and averaged to create a scale score.
Family Conflict | 6-week
  5-item measure from the Family, Friends and Self (FFS) assessment scales (Simpson & McBride, 1992; Hispanic Journal of Behavioral Sciences, 14, 327-340). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.
Family Communication | 6-week
  10-item measure assessing open vs. problem communication (McCubbin, Thompson & McCubbin, 1996; Family assessment: Resiliency, coping and adaptation - Inventories for research and practice. Madison, WI: University of Wisconsin). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.
Parent Support | 6-week
  4-item measure (Wills et al., 2004; Psychology of Addictive Behaviors, 18, 122-134). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.
Positive Family Relations | 12-week
  6-item Positive Family Relations measure adapted from the Cohesion subscale of Moos & Moos Family Environment Scale (Metzler et al., 1998; Journal of Family Psychology, 12, 600-619). Items are rated on a 5-point scale ("not at all" to "very much") and averaged to create a scale score.
Family Conflict | 12-week
  5-item measure from the Family, Friends and Self (FFS) assessment scales (Simpson & McBride, 1992; Hispanic Journal of Behavioral Sciences, 14, 327-340). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.
Family Communication | 12-week
  10-item measure assessing open vs. problem communication (McCubbin, Thompson & McCubbin, 1996; Family assessment: Resiliency, coping and adaptation - Inventories for research and practice. Madison, WI: University of Wisconsin). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.
Parent Support | 12-week
  4-item measure (Wills et al., 2004; Psychology of Addictive Behaviors, 18, 122-134). Items are rated on a 5-point scale ("never" to "almost always") and averaged to create a scale score.

SECONDARY OUTCOMES:
Lifetime and Past Month Substance Use | 6-week
  Number of times used in lifetime (range: "0 times" to "7 or more times") and number of days used in past month (range: "0 days" to "20-30-days") for each of the following substances: cigarettes; alcohol; marijuana; inhalants; any other illegal drug or pill to get high; over-the-counter medicines or OTCs to get high; and prescription medicines to get high.
  Additional items ask about quantity of cigarette, alcohol and marijuana use on days used, as well as intentions to use each of these substances in next 6 months (4-point scale, ranging from "definitely yes" to "definitely no").
Academic Performance | 6-week
  Items ask about typical grades in past month (range: "mostly A's" to "mostly F's"), school attachment (4-item measure from National Longitudinal Study of Adolescent Health), highest level of school the youth plans to finish (range: "I may not finish high school" to "I plan to go to graduate or professional school"), number of days skipped school in past month, and history of suspension from school.
Delinquency | 6-weeks
  13-item measure that includes items from Project ALERT and National Longitudinal Study of Adolescent Health. Items are rated on a 7-point scale ("0 days" to "20-30 days").
Lifetime and Past Month Substance Use | 12-week
  Number of times used in lifetime (range: "0 times" to "7 or more times") and number of days used in past month (range: "0 days" to "20-30-days") for each of the following substances: cigarettes; alcohol; marijuana; inhalants; any other illegal drug or pill to get high; over-the-counter medicines or OTCs to get high; and prescription medicines to get high.
  Additional items ask about quantity of cigarette, alcohol and marijuana use on days used, as well as intentions to use each of these substances in next 6 months (4-point scale, ranging from "definitely yes" to "definitely no").
Academic Performance | 12-week
  Items ask about typical grades in past month (range: "mostly A's" to "mostly F's"), school attachment (4-item measure from National Longitudinal Study of Adolescent Health), highest level of school the youth plans to finish (range: "I may not finish high school" to "I plan to go to graduate or professional school"), number of days skipped school in past month, and history of suspension from school.
Delinquency | 12-weeks
  13-item measure that includes items from Project ALERT and National Longitudinal Study of Adolescent Health. Items are rated on a 7-point scale ("0 days" to "20-30 days").

CONTACTS AND LOCATIONS:
Overall Officials: Joan S. Tucker, PhD, Principal Investigator — RAND
Locations (1):
- Centinela Youth Services, Hawthorne, California, United States